CLINICAL TRIAL: NCT01587547
Title: Amino Acid Profiling of Spent Culture Medium to Retrospectively Determine Individual Embryo Selection Criteria for Improved Clinical IVF Outcome
Brief Title: Amino Acid Profiling of Spent Culture Medium
Acronym: EmbryoSure
Status: Terminated | Type: Observational
Why Stopped: ORIGIO a/s acquired by Cooper Surgical Inc. who decided to withdraw from the project
Sponsor: Origio A/S (Industry)
Collaborators: Novocellus Ltd. (Unknown); Signifikans ApS (Other)
Responsible Party: Sponsor
Other Study IDs: DK005; CI/2010/0041 (Other: Medicines & Healthcare products Regulatory Agency (MHRA))
Record Dates: First submitted 2012-04-26; First posted 2012-04-30 (Estimated); Last update posted 2013-05-08 (Estimated); Status verified 2013-05

CONDITIONS: Infertility
Keywords: ART; IVF; ICSI; embryo selection
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Spent culture medium from the individual embryos
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- IVF and ICSI patients: Subjects undergoing IVF or ICSI treatment with a maximum of 2 embryos transferred

SUMMARY:
The purpose of this study is to develop an algorithm for embryo selection based on amino acid profiling (AAP) of spent culture medium. Development of the algorithm will be based on the ongoing implantation rate of the individual embryos transferred. As evaluated by ultrasound scan in gestational week 7.

DETAILED DESCRIPTION:
IVF/ICSI treatment has permitted many thousands of couples to conceive worldwide yet is limited by low success rates (in UK, approx. 25% live birth rate/treatment cycle for women up to 42 years of age; HFEA Annual Report, 2006) and a confounding high multiple birth rate (23%) due to the transfer of more than a single pre-implantation embryo. Multiple births are associated with prematurity, increased neonatal and maternal mortality and child handicap as well as being a major burden for health care systems. These problems have been highlighted in the data published by the HFEA (2009), which has called for "a professionally-led, coordinated national strategy to reduce the number of multiple births". This challenge could be met if single embryos of known developmental competence could be selected for transfer, thereby making the embryo selection process even more crucial. However, current non-invasive embryo selection criteria using light microscope analysis have limited predictive value for ongoing pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Minimum 4 x 2PN´s on Day 1 post insemination
* Subjects undergoing IVF or ICSI treatment with a maximum of 2 embryos transferred
* Both partners should be capable of understanding the study to which they are consenting
* Females > 18 and ≤ 40 years of age
* Regular menstrual cycle 21-35 days (both inclusive)
* Women treated with a standard drug protocol

Exclusion Criteria:

* The couple has previously participated in the DK005 study
* Use of assisted hatching
* Indication for TESA or PESA
* Any medical conditions or genetic disorders prohibiting IVF/ICSI or interfering with the interpretation of results of the study (including pre- implantation genetic diagnostics).
* Use of any investigational drug within 30 days before oocyte retrieval
* Any severe chronic disease of relevance for reproductive function.
* Oocyte donation patients (donor or recipient).

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Subjects will be recruited from couples and single women attending the IVF clinic for IVF/ICSI treatment.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2012-04; Primary Completion 2012-12 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Amino acid profile | After 24 hours of culture
  Amino acid profiling (AAP) will be performed of spent culture medium from individually cultured embryos. AAP results will be correlated to the ongoing implantation rate week 7 as well as morphological embryo development parametres.

SECONDARY OUTCOMES:
Ongoing clinical pregnancy rate | Gestational week 7
  Evaluated by ultrasound scan

CONTACTS AND LOCATIONS:
Overall Officials: Helen M Picton, BSc, PhD, Principal Investigator — Leeds Institute of Genetic Health
Locations (2):
- United Kingdom (2):
  - The Hewitt Centre for Reproductive Medicine, Liverpool Women's Hospital, Liverpool
  - Hammersmith IVF, Hammersmith Hospital, London